CLINICAL TRIAL: NCT05582590
Title: A Phase 1 Open-Label Dose-Escalation Study of the Safety of Adoptively Transferred Autologous CD8+ T Lymphocytes Targeting HPV-16 E6/E7, HPV-18 E6/E7 and Survivin in Patients With Relapsed or Refractory HPV-related Oropharyngeal Cancers
Brief Title: Autologous T Cells Targeting HPV16 HPV18 & Survivin in Patients With R/R HPV-related Oropharyngeal Cancers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NexImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEXI-003-HPV-101
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Oropharyngeal Cancer; Human Papilloma Virus; Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma; Oropharyngeal Cancer, Metastatic; Head and Neck Cancer Metastatic; HPV-Related Squamous Cell Carcinoma; HPV-Related Mucosal Head and Neck Squamous Cell Carcinoma; Relapsed Oropharyngeal SCC; Refractory Oropharyngeal Squamous Cell Carcinoma
Keywords: relapsed or refractory HPV-related oropharyngeal cancer; human papilloma virus-related cancer; HPV-related head and neck cancer; HPV-related oropharyngeal cancer; cell therapy; adoptive cell therapy; NEXI-003; Head and neck cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Recurrence | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Standard 3+3 study design for the Dose Escalation Stage and a Dose Expansion Stage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): 2 x 10^8 NEXI-003 T cells (derived from peripheral blood mononuclear cells [PBMCs] of the patient) administered by intravenous infusion on Day 1 of each cycle
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: NEXI-003 T cells
- Cohort 2 (Experimental): 2 x 10^8 NEXI-003 T cells (derived from peripheral blood mononuclear cells [PBMCs] of the patient) administered by intravenous infusion on Days 1 and 8 of each cycle
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: NEXI-003 T cells
- Cohort 3 (Experimental): 2 x 10^8 NEXI-003 T cells (derived from peripheral blood mononuclear cells [PBMCs] of the patient) administered by intravenous infusion on Days 1, 8, and 15 of each cycle
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: NEXI-003 T cells
- Cohort 4 (Experimental): 4 x 10^8 NEXI-003 T cells (derived from peripheral blood mononuclear cells [PBMCs] of the patient) administered by intravenous infusion on Day 1, and 2 x 10^8 NEXI-003 T cells administered by intravenous infusion on Days 8 and 15 of each cycle
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: NEXI-003 T cells
- Dose Expansion Stage (Experimental): Dose Expansion Stage to further define the safety and clinical activity, and to confirm the recommended Phase 2 dose of the NEXI- 003 T cell product at the dose established from the Dose Escalation Stage.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: NEXI-003 T cells

INTERVENTIONS:
Drug: Fludarabine — Lymphodepletion Chemotherapy on Days -5, -4, and -3 before Cycle 1 ONLY
  Other Names: Fludara
Drug: Cyclophosphamide — Lymphodepletion Chemotherapy administered on Days -5, -4, and -3 before Cycle 1 ONLY
  Other Names: Cytoxan
Biological: NEXI-003 T cells — Adoptive Cell Therapy specified dose on specified day(s)

SUMMARY:
This is a multicenter, open-label, Phase I, first-in-human trial to characterize the safety and clinical activity of an antigen-specific CD8+ T-cell product in patients with relapsed or refractory locally advanced or metastatic HPV-related oropharyngeal cancers. Patients must have received at least one prior standard treatment regimen consisting of systemic immunotherapy and/or chemotherapy. The investigative agent is an autologous adoptive T-cell product derived from the patient's endogenous cytolytic T cells that are directed toward HPV-16 E6/E7, HPV-18 E6/E7 antigens, and a tumor-associated antigen (Survivin) by ex vivo exposure to an artificial antigen presenting cell to which HLA-A2 antigen-peptides have been fit within the pocket of an MHC class 1 molecule. Patients must express HLA-A*0201.

DETAILED DESCRIPTION:
The primary objective is to assess the safety of NEXI-003 in patients with relapsed or refractory HPV-related oropharyngeal cancers. The study will consist of two stages: a Dose-Escalation (Stage 1) and a Dose Expansion (Stage 2).

The first stage of the trial is the Dose-Escalation (Stage 1). A standard dose-escalation 3+3 design will be utilized to identify a safe maximum tolerated dose (MTD) of NEXI-003 in patients with relapsed or refractory HPV-related oropharyngeal cancers. The MTD of NEXI-003 T cells will be identified during the first 28-day cycle (Cycle 1) of the Dose-Escalation Stage, which is defined as the DLT period. A total of 4 dosing cohorts are planned in the Dose Escalation Stage.

Initially 3 patients are enrolled into a dosing cohort. After all 3 patients in a cohort have been followed for 28 days of Cycle 1 (the DLT Period), the safety information will be assessed by the Data Review Committee (DRC). If no DLT is reported in the first 3 patients enrolled during the 28-day initial cycle of treatment (the DLT Period), enrollment into the next higher dose cohort may begin, after safety information is assessed by the DRC. If 1 of the first 3 patients has a DLT, then 3 more patients will be enrolled into that cohort. If a DLT occurs in ≥ 2 patients, then the MTD will be judged to have been exceeded and the next lower cohort dose will be considered the MTD. If a DLT occurs in ≤ 1 of 6 patients, then patients may be enrolled in the next highest dose level. The DRC will review eligibility criteria, doses of all study treatments and safety data and make recommendations as to the further conduct of the study. If ≥ 2 patients in Cohort 1 experience a DLT, then Cohort -1 (1 x 10^8 NEXI-003 T cells on Day 1 of Cycle 1; stepdown dose, if needed) will be evaluated using the 3+3 design.

After identification of the MTD, or the finding that the last dosing cohort is tolerated well (i.e., the maximum practical dose [MPD]), 12 patients will be enrolled to receive NEXI-003 treatment at the MTD/MPD level in the Dose Expansion Stage to gain additional safety, clinical activity, and pharmacokinetic data (i.e., persistence and expansion) of the NEXI-003 antigen specific CD8+ T cell product. Safety, clinical activity, and pharmacokinetic data from the Dose Escalation and Dose Expansion stages will be assessed to determine the recommended Phase 2 dose (RP2D).

Patients in both the Dose Escalation and Dose Expansion Stages may receive additional cycles of NEXI-003 per investigator discretion and if protocol-specified criteria are met.

Each of the two stages of the study will consist of the following three consecutive study periods for each patient: Pretreatment Period (consisting of Screening, Leukapheresis/Manufacturing, and Baseline Re-evaluation), Treatment Period (consisting of lymphodepletion [LD] chemotherapy and NEXI-003 treatment), and Post-Treatment Period (consisting of Post-treatment Follow-up and Survival Follow-up). The Pretreatment Period will be approximately 4 to 6 weeks. The Treatment Period will consist of at least 28-day cycle (i.e., 4 weeks), and per investigator discretion if the patient meets protocol-specified criteria, the patient may receive additional 4-week cycles. The Post-Treatment Follow-up Period will consist of up to 9 months of post-treatment assessments, and up to 9 months of survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. The patient will be typed for HLA-A*0201 expression as determined by high resolution sequence-based typing method. If documented HLA results are available from a previous test, the patient can be enrolled using these results after review and approval by the sponsor.
2. Patients with cytologically or histologically confirmed locally advanced or metastatic HPV related oropharyngeal cancers with confirmed detection of HPV-16 and/or HPV-18.
3. Patients with HPV-related oropharyngeal cancers who have received at least 1 prior line of standard-of-care (SOC) treatment (for example, per the current NCCN Guidelines for Patients with Oropharyngeal Cancer) consisting of systemic immunotherapy and/or chemotherapeutic treatment.

   1. The last dose of cytotoxic chemotherapy and/or steroids must be administered at least 28 days prior to the leukapheresis procedure.
   2. Any adverse event(s) that the patient may have experienced from prior therapy must have resolved to ≤ Grade 1 according to NCI CTCAE version 5.0.
4. Measurable disease per RECIST v1.1 criteria (at least 1 lesion that can be measured accurately in at least 1 dimension with the longest diameter ≥ 10 mm [MRI or CT scan sliced thickness ≤ 5 mm]).
5. Pulse oximetry ≥ 92% on room air.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Life expectancy of at least 3 months.
8. Be willing to comply with the study schedule and all other protocol requirements.
9. Women of childbearing potential (WOCBP), defined as a sexually mature woman who has not undergone a hysterectomy or tubal ligation or who has not been naturally postmenopausal for at least 24 consecutive months, must have 2 negative pregnancy tests prior to treatment. All sexually active WOCBP and all sexually active male patients must agree to use highly effective methods of birth control throughout the study.
10. Ability of the patient to understand and willingness to sign a written informed consent form.

Exclusion Criteria:

1. A diagnosis of other malignancies if the malignancy has required therapy within the last 3 years or is not in complete remission. Exceptions are non-metastatic basal cell or squamous cell carcinomas of the skin or prostate cancer that does not require treatment. Patients taking adjuvant hormonal therapy for definitively treated cancers (e.g., breast cancer, prostate cancer) are eligible.
2. Major surgery within 28 days prior to the first study drug administration (minimally invasive procedures, such as diagnostic biopsies, are permitted).
3. Known central nervous system involvement.
4. Treatment with an allogeneic hematopoietic stem cell transplantation.
5. Treatment with any investigational agent(s) at the time of informed consent.
6. Left ventricular ejection fraction (LVEF) < 45%, congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), unstable angina, serious uncontrolled cardiac arrhythmia, a myocardial infarction within 6 months prior to study entry or a history of myocarditis.
7. The following hematological laboratory results at Screening (these results must be independent of blood product or hematopoietic growth factor support):

   1. Hemoglobin < 9.0 g/dL.
   2. Platelet count < 100,000/μL.
   3. Absolute neutrophil count (ANC) < 1000/ μL.
8. The following chemistry laboratory results at Screening:

   1. Serum creatinine ≥ 1.5 mg/dL or estimated glomerular filtration rate (eGFR) ≤ 50 mL/min/1.73 m^2.
   2. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3x the upper limit of normal (ULN) or serum total bilirubin > 2 mg/dL (except for patients in whom hyperbilirubinemia is attributed to Gilbert's Syndrome).
9. International normalized ratio (INR) or activated partial thromboplastin time (aPTT) > 1.5x ULN within 1 week prior to the start of lymphodepletion chemotherapy, unless on a stable dose of an anticoagulant.
10. Are pregnant or breastfeeding.
11. Vaccination with any live virus vaccine is not permitted prior to the initiation of study treatment.

    1. Inactivated annual influenza vaccination is allowed.
    2. Vaccines such as COVID-19 vaccine, e.g., SARS-CoV-2 vaccine > 7 days before administration is acceptable. For vaccines requiring more than 1 dose, the full regimen should be completed prior to Cycle 1 Day 1.
12. Active bacterial, viral, or fungal infection within 72 hours of the start of lymphodepletion chemotherapy; patients with ongoing use of prophylactic antibiotics, antifungal agents, or antiviral agents remain eligible as long as there is no evidence of active infection.
13. Have human immunodeficiency virus (HIV) active infection as indicated by positive HIV polymerase chain reaction (PCR) test, human T-cell leukemia virus type 1 infection, or hepatitis B virus (HBV) or hepatitis C virus (HCV) viremia or are at risk for HBV reactivation (at risk for HBV reactivation is defined as being hepatitis B surface antigen [HbsAg] positive, or anti-HBe-antibody positive), or are positive for HBV DNA. HCV ribonucleic acid (RNA) must be undetectable by laboratory test.
14. Any condition including the presence of laboratory abnormalities, that places the patient at an unacceptable risk if the patient was to participate in the study.
15. Have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).

    Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is permitted.
16. Patients who experienced the following immune checkpoint inhibitor-related AEs even if the AE resolved to ≤ Grade 1 or baseline:

    1. ≥ Grade 3 ocular AE
    2. Changes in liver function tests that met the criteria for Hy's Law (> 3× ULN of either ALT/AST with concurrent > 2× ULN of total bilirubin (total and direct) and without alternate etiology)
    3. ≥ Grade 3 neurologic toxicity
    4. ≥ Grade 3 colitis
    5. ≥ Grade 3 renal toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 12 months
  Frequencies of patients with treatment-emergent AEs (TEAEs)
Dose-Limiting Toxicities (DLTs) | 28 days
  DLTs in Cycle 1
Severities of AEs | 12 months
  Frequencies of patients with treatment-emergent AEs (TEAEs) by severity
Relationship of AEs | 12 months
  Frequencies of patients with treatment-emergent AEs (TEAEs) by relationship to NEXI-003 T cells
Serious Adverse Events (SAEs) | 12 months
  Frequencies of patients with treatment-emergent SAEs
Adverse Events of Special Interest (AESIs) - Cytokine Release Syndrome (CRS) | 12 months
  Frequencies of patients with treatment-emergent CRS
Adverse Events of Special Interest (AESIs) - Immune Effector cell-associated neurotoxicity syndrome (ICANS) | 12 months
  Frequencies of patients with treatment-emergent ICANS

SECONDARY OUTCOMES:
Overall response rate (ORR) | 12 months
  ORR as measured by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1
Duration of response (DoR) | 12 months
  Response as measured by RECIST v1.1 over time
Determine the persistence of NEXI-003 T cells in peripheral blood | 12 months
  Determine NEXI-003 at pre-dose and different times post-dose by multimer-based staining of antigen-specific NEXI-003 T cells.
Determine manufacturing feasibility by assessing the manufactured product for Cell Viability | 1 month
  Percent NEXI-003 T cell viability in each manufactured product
Determine manufacturing feasibility by assessing the manufactured product for Cell Yield | 1 month
  Total cell count for each manufactured product
Determine manufacturing feasibility by assessing the manufactured product for Percent CD3+/CD4- T cells | 1 month
  Percent of CD3+/CD4- T cells in each NEXI-003 T cell product
Determine manufacturing feasibility by assessing the manufactured product for Percent CD3+/CD8+ T cells | 1 month
  Percent of CD3+/CD8+ T cells in each NEXI-003 T cell product
Determine manufacturing feasibility by assessing the memory immunophenotypes in the manufactured product | 1 month
  Percent of antigen-specific-NEXI-003 T cell memory immunophenotypes in the investigational product